CLINICAL TRIAL: NCT00444782
Title: "Heptovax" - A Phase II, Open-Label Trial Evaluating the Safety and Efficacy of GV1001 in Advanced Hepatocellular Carcinoma.
Brief Title: A Phase II, Open-Label Trial Evaluating GV1001 in Advanced Hepatocellular Carcinoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmexa A/S (Industry)
Responsible Party: Lotte Rosendahl, Pharmexa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX115.1.1-201
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Advanced Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — GV1001 peptide

INTERVENTIONS:
Biological: GV1001

SUMMARY:
The purpose of this study is to investigate the efficacy of GV1001 in locally advanced or metastatic HCC. Also the safety of GV1001 and immunogenicity will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma diagnosis fulfilling one of the following criteria (as per the American Association for the Study of Liver Diseases [AASLD] guidelines, see Appendix 5):

  1. Nodule in a cirrhotic or non-cirrhotic liver with a biopsy showing HCC;
  2. Nodule in cirrhotic liver where no biopsy is performed:

     * Nodules between 1-2 cm in a cirrhotic liver with a typical coincidal vascular pattern of HCC (i.e. hypervascular with washout in the portal/venous phase) in two dynamic studies: either CT scan, contrast ultrasound or MRI with contrast.
     * Nodule larger than 2 cm in a cirrhotic liver with a typical vascular pattern of HCC on a dynamic imaging technique.

Please note: HCC in a non-cirrhotic liver can only be diagnosed with a biopsy showing HCC.

* Measurable disease according to modified RECIST (see Appendix 7).
* At least one treatment-naïve target lesion (treatment-naïve being defined as not having been treated with local therapy, such as surgery, radiation therapy, hepatic arterial embolisation, chemoembolisation, radio-frequency ablation or cryo-ablation).
* Barcelona Clinic Liver Cancer (BCLC) stage A, B or C (see Appendix 6) (Stage D is excluded).
* Child-Pugh stage A (see Appendix 8).
* Male or female aged 18 years or older.
* Adequate haematological parameters, as demonstrated by:

  * Haemoglobin greater than or equal to 9.0 g/dL (SI units: 5.6 mmol/L);
  * WBC greater than or equal to 3.0 x 109/L;
  * Platelets greater than or equal to 75 x 109/L.
* ALT and AST ≤ 5 times the upper limit of normal.
* Bilirubin < 2 mg/dL.
* Serum creatinine smaller than or equal to 1.5 mg/dL (SI units: 132 µmol/L).
* Performance status ECOG 0 or 1.
* Minimum life expectancy of 3 months at screening.
* Written informed consent given prior to any study specific procedures.

Exclusion Criteria:

* HCC amenable to curative treatment or transplantation.
* History of other malignancies in the last 5 years (10 years in the case of breast cancer), except for adequately treated non-melanoma skin cancers (Basal Cell Carcinoma, Squamous Cell Carcinoma) and carcinoma in situ of the cervix.
* Known history of or co-existing autoimmune disease.
* Known Central Nervous System (CNS) metastases.
* Known history of human immunodeficiency virus (HIV).
* Any medical condition that, in the opinion of the Investigator, may compromise the compliance of the patient to receive study treatment and follow study procedures.
* Treatment with any other IMP within 4 weeks prior to cyclophosphamide administration at Day -3.
* Known sensitivity to any components of cyclophosphamide, GV1001 or GM-CSF.
* Concomitant treatment with the following within 4 weeks of pre-treatment with cyclophosphamide:

  * Anti-tumour treatment (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, cytokines, interferons, protease inhibitors, and gene therapy) and vaccines.
  * Chronic corticosteroids (inhaled and topical steroids are permitted including low dose steroids at non-immunosuppressive doses e.g. 15 mg prednisolone daily for up to 7 days).
  * Herbal medicine either containing hypericum perforacum (e.g., St Johns Wort) or claiming to have anti-tumour effects (e.g., Iscador).
* Pregnancy or lactation.
* Women of childbearing potential not using reliable and adequate contraceptive methods, defined as the use of oral, implanted, injectable, mechanical or barrier products for the prevention of pregnancy; or women who are practising abstinence; or where the partner is sterile, for example a vasectomy.
* Unable for any other reason to comply with the protocol (treatment or assessments).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Response rate (Partial and Complete Response) according to modified RECIST.

SECONDARY OUTCOMES:
Time to Progression (TTP)
Time to Symptomatic Progression (TTSP)
Progression Free Survival (PFS)
Immune Response

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Rosendahl, Pharmacist (CTM), Study Chair — Pharmexa A/S
Locations (3):
- Michel Beaugrand, Bondy, France
- Tim F. Greten, Hanover, Germany
- Jordi Bruix, Barcelona, Spain

REFERENCES:
- [Derived] Greten TF, Forner A, Korangy F, N'Kontchou G, Barget N, Ayuso C, Ormandy LA, Manns MP, Beaugrand M, Bruix J. A phase II open label trial evaluating safety and efficacy of a telomerase peptide vaccination in patients with advanced hepatocellular carcinoma. BMC Cancer. 2010 May 17;10:209. doi: 10.1186/1471-2407-10-209. PMID 20478057